CLINICAL TRIAL: NCT04293003
Title: Short-term Metabolic Effects of Morning Energy Restriction Versus Two Different Early-day Nutrition Strategies
Brief Title: Metabolic Effects of Morning 16/8 Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 39/12-02-2019
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting (Experimental): 6-hour morning fasting
  Interventions: Other: fasting
- Low carbohydrate (Experimental): Consumption of a zero-carbohydrate breakfast
  Interventions: Other: Low carbohydrate
- Mediterranean (Experimental): Consumption of a Mediterranean breakfast
  Interventions: Other: Mediterranean

INTERVENTIONS:
Other: fasting — 6-hour fasting
  Arms: Fasting
Other: Low carbohydrate — Consumption of a zero-carbohydrate breakfast
  Arms: Low carbohydrate
Other: Mediterranean — Consumption of a Mediterranean-type breakfast
  Arms: Mediterranean

SUMMARY:
A study to address the effects of early-day fasting on fat tissue mobilization in comparison to a typical isocaloric Mediterranean and a low-carbohydrate breakfast.

DETAILED DESCRIPTION:
The study design meets a cross-over pattern with 3 different morning visits of 6 hour duration each. After an informed consent is received from the participant, a crude medical history, physical examination and collection of somatometric data through bio-impendance analysis will take place. An intravenous catheter will be placed in the participants forearm.

At zero time point, depending on study visit, participants will either (A) remain fasted (B) start consuming ta pre-prepared zero-carbohydrate 500 kcal test meal (C) start consuming ta pre-prepared 500 kcal test meal with a composition conforming to a standard Mediterannean breakfast. Participants will be given 10 minutes to consume the meal.

Blood samples will be drawn and visual analogue scales (VAS) for hunger and satiety will be filled in at the following time points (min): -15, 0, 15, 30, 60, 90, 120, 180, 240, 300, 360.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25 kg/m2
* Willfulness to participate

Exclusion Criteria:

* Overweight or obesity (BMI>25 kg/m2)
* Type 1 or 2 diabetes mellitus
* Uncontrolled thyroid disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Mobilisation of adipose tissue | 6 hours
  Area Under the Curve (AUC) of free fatty acid (FFA) and beta-Hydroxybutyrate (bOB) concentration

SECONDARY OUTCOMES:
Mobilisation of gut peptides | 6 hours
  AUC of Ghrelin, Peptide YY and glucagon-like peptide -1 (GLP-1) concentration
Degree of appetite suppression | 6 hours
  Visual Analogue Scale score (0-10, 0 equals minimal and 10 equals highest) for appetite
Degree of satiety induction | 6 hours
  Visual Analogue Scale score (0-10, 0 equals minimal and 10 equals highest) for satiety

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No